CLINICAL TRIAL: NCT01475695
Title: An Open Label, Non-Randomized, Single Dose, Mass Balance Study to Investigate the Recovery, Excretion, and Pharmacokinetics of 14C-GSK2251052 Administered as a Single Intravenous Dose to Healthy Adult Subjects
Brief Title: GSK2251052 Mass Balance in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 115243
Record Dates: First submitted 2011-11-17; First posted 2011-11-21 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Community-acquired Infection
Keywords: Mass balance; intravenous; GSK2251052; Healthy volunteer; Antimicrobial; Radiolabel
MeSH Terms: conditions — Community-Acquired Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single cohort (Experimental): 14C GSK2251052
  Interventions: Drug: 14C GSK2251052

INTERVENTIONS:
Drug: 14C GSK2251052 — 1500 mg iv dose GSK2251052

SUMMARY:
Approximately 6 healthy male subjects will be administered a single 1500 mg intravenous dose of 14C-GSK2251052 under fasted conditions. Blood, urine and fecal samples will be collected for a minimum of 14 days following study drug administration. Safety and tolerability will be monitored throughout the study. A follow-up visit will occur 7-14 days after study drug administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and ECG. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male between 30 and 55 years of age inclusive, at the time of signing the informed consent.
* Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication through at least 90 days following the dose of GSK2251052.
* Body weight equal to or greater than 50 kg and BMI within the range 18.5-30.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* QTcB less than 450 msec or QTc less than 480 msec in subjects with Bundle Branch Block.
* Available to complete the study and return for follow-up visits if necessary.
* A history of regular bowel movements (averaging one or more bowel movements per day).
* AST, ALT, alkaline phosphatase and bilirubin equal to or less than 1.5xULN (isolated bilirubin greater than 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35%).

Exclusion Criteria:

* Female subjects.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of greater than 21 units for males or greater than14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (approximately 240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice [and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices] from 7 days prior to the first dose of study medication.
* Subjects who have received a total body radiation dose of greater than 5.0 mSv (upper limit of WHO category II) or exposure to significant radiation (e.g. serial x-ray or CT scans, barium meal etc) in the 12 months prior to this study.
* Any condition that could interfere with the accurate assessment and recovery of radioactivity [14C].
* Participation in a clinical trial involving administration of 14C-labelled compound(s) within the last 12 months.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy should be excluded.
* The subject's systolic blood pressure is outside the range of 90-140 mmHg, or diastolic blood pressure is outside the range of 45-90 mmHg or heart rate is outside the range of 45-100 bpm. A single repeat is allowed to determine eligibility.
* Exclusion criteria for screening ECG per protocol.(a single repeat is allowed for eligibility determination).

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-04-21 (Actual); Primary Completion 2011-05-19 (Actual); Study Completion 2011-05-19 (Actual)

PRIMARY OUTCOMES:
Evaluate pharmacokinetic parameters for GSK2251052 and radiolabeled compound following intravenous dose | Up to 14 days
Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time | Up to 14 days
Area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration within a subject across all treatments | Up to 14 days
Maximum observed concentration | Up to 14 days
Time of occurrence of maximum observed concentration | Up to 14 days
Terminal phase half-life | Up tp 14 days
Systemic clearance of parent drug | Up to 14 days
Volume of distribution | Up to 14 days
Percent recovery of total radiocarbon in urine and feces | Up to 14 days
Urine, fecal recovery and total recovery of radioactivity (as a percentage of total radioactive dose in each interval and cumulative) | Up to 14 days

SECONDARY OUTCOMES:
Adverse events, vital signs, electrocardiogram and clinical laboratory assessments. | Up to 14 days
Collection of samples for characterization and quantification, or estimation, of GSK2251052-related metabolites in plasma, urine and fecal homogenates to be conducted under a separate protocol. | Up to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Zuidlaren, Netherlands

REFERENCES:
- [Background] Bowers GD, Tenero D, Patel P, Huynh P, Sigafoos J, O'Mara K, Young GC, Dumont E, Cunningham E, Kurtinecz M, Stump P, Conde JJ, Chism JP, Reese MJ, Yueh YL, Tomayko JF. Disposition and metabolism of GSK2251052 in humans: a novel boron-containing antibiotic. Drug Metab Dispos. 2013 May;41(5):1070-81. doi: 10.1124/dmd.112.050153. Epub 2013 Feb 25. PMID 23439661
- See also: Results for study 115243 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/115243?search=study&search_terms=115243#rs